CLINICAL TRIAL: NCT06243341
Title: The Impact of Lepidium Meyenii (MACA) Supplementation on Basketball-related Performance and Anti-fatigue Ability: a Double Blind Crossover Study
Brief Title: The Impact of MACA Supplementation on Basketball-related Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 113-1
Record Dates: First submitted 2024-01-14; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Sports
Keywords: Lepidium meyenii; Basketball Jump Shooting Accuracy Test; Repeated Sprint Ability Test; blood lactate clearance rate; ergogenic aids

STUDY DESIGN:
Intervention Model Description: a double blind crossover study
Who Masked: Investigator
Masking Description: a double blind crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MACA (MC) (Experimental): Daily MACA supplementation for two weeks.
  Interventions: Dietary Supplement: Lepidium meyenii (MACA)
- placebo (Placebo Comparator): Daily placebo supplementation for two weeks.
  Interventions: Dietary Supplement: Lepidium meyenii (MACA)

INTERVENTIONS:
Dietary Supplement: Lepidium meyenii (MACA) — The MACA supplement is derived from a concentrated 6:1 blend of black, red, and yellow MACA root compounds, with an 80:15:5 ratio respectively.
  Other Names: 100% corn-starch maltodextrin powder

SUMMARY:
In this randomized crossover study, ten elite healthy male basketball players were included. Following a 17:00 PM training routine, participants completed a two-week supplementation with 2000 mg of MACA or placebo. After supplementation, participants underwent a Basketball Jump Shooting Accuracy Test and Repeated Sprint Ability Test.

DETAILED DESCRIPTION:
Supplementation with Lepidium meyenii (MACA) has been shown in animal studies to increase blood lactate clearance and rapid lactate removal, which may be effective in reducing fatigue during intermittent exercise. However, no studies have investigated the effects of MACA supplementation on interval exercise and basketball performance. We hypothesized that MACA supplementation could reduce fatigue and improve performance in elite healthy male basketball players. This study aimed to determine the effectiveness of MACA compared to placebo on overall basketball performance.

ELIGIBILITY:
Inclusion Criteria:

* (i) healthy male adults, those individuals who are free of pain, insomnia, or other injuries recently, without any medication used in recent 2 months,
* (ii) basketball players competing in a Taiwan university basketball association for more than two years.

Exclusion Criteria:

* (i) were below 20 years old,
* (ii) did not have won at least eighth place in national-level basketball competitions,
* (iii) were with cardiovascular diseases or any disease that made subjects feel ill.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only adult male participants were recruited
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Countermovement jump test | immediately after 2 weeks intervention
  Three jumps were measured with 1 minute rest for each participant.

SECONDARY OUTCOMES:
Basketball Jump Shooting Accuracy Test | immediately after 2 weeks intervention
  The first test was the basketball jump shooting Accuracy Test (BJSAT), which has been used in the past with sufficient reliability to two and three-point shooting accuracy
Repeated Sprint Ability Test | immediately after 2 weeks intervention
  Repeated Sprint Ability test (40× 15m with a 1:4, exercise : rest time ratio, such as 2 seconds :8 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Che-Hsiu Chen, PhD, Study Director — Sport Science Research Center
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No personal data of participants will be provided

REFERENCES:
- [Result] Stone M, Ibarra A, Roller M, Zangara A, Stevenson E. A pilot investigation into the effect of maca supplementation on physical activity and sexual desire in sportsmen. J Ethnopharmacol. 2009 Dec 10;126(3):574-6. doi: 10.1016/j.jep.2009.09.012. Epub 2009 Sep 23. PMID 19781622
- [Derived] Wu PS, Wu SH, Jiang RS, Chen CH, Chen BW, Chiu CH. The Impact of Lepidium meyenii (MACA) Supplementation on Basketball-related Performance and Antifatigue Ability: A Double-blind Crossover Study. J Physiol Investig. 2025 Sep 1;68(5):297-304. doi: 10.4103/ejpi.EJPI-D-25-00037. Epub 2025 Sep 17. PMID 40960048

DOCUMENTS (1):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT06243341/Prot_000.pdf